CLINICAL TRIAL: NCT00505557
Title: Dual-Plane Breast Augmentation: Axillary Approach With Assistant of Endoscope
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chinese Academy of Sciences (Other Government)
Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 621125-1
Record Dates: First submitted 2007-07-20; First posted 2007-07-23 (Estimated); Last update posted 2009-06-24 (Estimated); Status verified 2009-06

CONDITIONS: Mammoplasty
Keywords: augmentation mammoplasty; Dual plane; Endoscope; Transaxillary incision

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Transaxillary dual plane technique

SUMMARY:
The purpose of this study is to evaluate the feasibility and outcome of performing dual plane breast augmentation with assistant of endoscope by axillary approach.

DETAILED DESCRIPTION:
Dual plane augmentation mammoplasty is a logical approach to realize the benefits of retromammary and partial retropectoral implant placement while minimizing the tradeoffs of other pocket locations. Traditionally, dual plane augmentation has been performed using transareolar or inframammary fold approach. However, the approach is unacceptable to Chinese patients because of the front scar formation. For aesthetic reasons, the axillary incision is more acceptable approach for augmentation mammoplasty.

The endoscope assistant technique has been widely used in transaxillary breast augmentation. It provides the feasibility to perform dual plane breast augmentation by axillary approach.

In this research, at least 40 patients with light degree of glandular ptotic and constricted lower pole breasts are selected to receive soft cohesive gel microtextured anatomic style silicone implants. Portions of the pectoralis major muscle is split without its release from the costal margin with the help of a 10mm, 30°endoscope and endoscopic diathermy scissors through a 4-cm incision in the axilla each side. Bleeding during surgery is kept to the minimum. The results of outcomes, operative time, bleeding volume, drainage volume, complications are observed.

ELIGIBILITY:
Inclusion Criteria:

* All women who want breast augmentation using the implants.Especially for the patients with
* glandular ptotic (< I degree) breasts
* thick soft tissues (> 10 mm) in the low pole of the breast

Exclusion Criteria:

* With thin soft tissues (< 9 mm) in the low pole of the breast

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2006-05; Primary Completion 2007-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
98% of the patient satisfied with softer, more natural breasts. The procedure provided more accurate bleeding control, faster postoperative coverage. | within half year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yilin Cao, M.D., Study Chair — Chinese Academy of Medical Sciences
Locations (1):
- Plastic Surgery Hospital Affilicated to Chinese Academy of Medical Sciences & Peking Union Medical College, Beijing, China

REFERENCES:
- [Background] Yu L, Wang J, Zhang B, Zhu C. Endoscopic transaxillary capsulectomy. Aesthetic Plast Surg. 2006 May-Jun;30(3):282-5. doi: 10.1007/s00266-005-0159-0. PMID 16733771
- [Background] Villafane O, Garcia-Tutor E, Taggart I. Endoscopic transaxillary subglandular breast augmentation using silicone gel textured implants. Aesthetic Plast Surg. 2000 May-Jun;24(3):212-5. doi: 10.1007/s002660010035. PMID 10890950
- [Background] Howard PS. The role of endoscopy and implant texture in transaxillary submuscular breast augmentation. Ann Plast Surg. 1999 Mar;42(3):245-8. doi: 10.1097/00000637-199903000-00003. PMID 10096613
- [Background] Howard PS, Oslin BD, Moore JR. Endoscopic transaxillary submuscular augmentation mammaplasty with textured saline breast implants. Ann Plast Surg. 1996 Jul;37(1):12-7. doi: 10.1097/00000637-199607000-00002. PMID 8826586
- [Background] Tebbetts JB. Dual plane breast augmentation: optimizing implant-soft-tissue relationships in a wide range of breast types. Plast Reconstr Surg. 2006 Dec;118(7 Suppl):81S-98S; discussion 99S-102S. doi: 10.1097/00006534-200612001-00012. PMID 17099485
- [Background] Tebbetts JB. Axillary endoscopic breast augmentation: processes derived from a 28-year experience to optimize outcomes. Plast Reconstr Surg. 2006 Dec;118(7 Suppl):53S-80S. doi: 10.1097/01.prs.0000247314.92351.99. PMID 17099484
- [Background] Tofield JJ. Dual plane breast augmentation. Plast Reconstr Surg. 2001 Dec;108(7):2162-4. doi: 10.1097/00006534-200112000-00069. No abstract available. PMID 11743433
- [Background] Tebbetts JB. Dual plane breast augmentation: optimizing implant-soft-tissue relationships in a wide range of breast types. Plast Reconstr Surg. 2001 Apr 15;107(5):1255-72. doi: 10.1097/00006534-200104150-00027. PMID 11373572